CLINICAL TRIAL: NCT02712697
Title: Treatment of Shentong Granules Plus Prednisone on Patients With Severe IgA Nephropathy(Ying-deficiency of the Liver and Kidney Pattern): a Randomized, Double-blind,Placebo-controlled Multicentre Clinical Trial
Brief Title: Integrative Medicine of IgA Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: RenJi Hospital (Other); Ruijin Hospital (Other); Shanghai 6th People's Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZY3- CCCX-2-1002
Record Dates: First submitted 2015-11-17; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2015-11

CONDITIONS: Primary IgA Nephropathy
Keywords: liver-kidney yin deficiency syndrome; primary severe IgA nephropathy; Lee's grade Ⅲ
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Hormones; Prednisone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- WM Group (Experimental): Shentong Granules, two packs, bid, P.O., 48weeks; Prednisone, 0.5-1mg/kg.d, P.O., eight to twelve weeks; then reduced to 30mg by reduce 5mg every two weeks; followed by the monthly reduction of 5mg, about 9-12 months
  Interventions: Drug: WM (Shentong Granules); Drug: Hormone (prednisone)
- Hormone Group (Placebo Comparator): Placebo ; Prednisone, 0.5-1mg/kg.d, P.O., eight to twelve weeks; then reduced to 30mg by reduce 5mg every two weeks; followed by the monthly reduction of 5mg, about 9-12 months
  Interventions: Drug: Hormone (prednisone)

INTERVENTIONS:
Drug: WM (Shentong Granules) — Shentong Granules with Prednisone
  Other Names: Shentong Granules
  Arms: WM Group
Drug: Hormone (prednisone) — Oral prednisone
  Other Names: prednisone

SUMMARY:
The present study was designed to identify the efficacy and safety of Integrative Medicine by joint oral steroid medicine on liver-kidney yin deficiency, severe IgA nephropathy. Furthermore, search for potential diagnostic predictor in IgA Nephropathy by Proteomics and Metabolomics.

DETAILED DESCRIPTION:
The present study was designed to identify the efficacy and safety of Integrative Medicine by joint oral steroid medicine on liver-kidney yin deficiency, severe IgA nephropathy. Furthermore, search for potential diagnostic predictor in IgA Nephropathy by Proteomics and Metabolomics. Combined with TCM Syndrome research, the investigators will clarify targets or mechanisms of herbal treatment. Eventually, to form a more clinically appropriate standardized combination treatment of severe IgA nephropathy.

ELIGIBILITY:
Inclusion Criteria:

1. The primary IgAN was confirmed by renal biopsy and clinical examination, and the pathological manifestations were Lee's grade and above;
2. TCM is liver kidney yin deficiency syndrome;
3. age 18-70 years old, sex, nationality is not limited;
4. CKD phase 2-4 （89 ml/min>eGFR（EPI Formula）>15ml/min/1.73m2）;
5. 24 hour urinary protein≥1g.

Exclusion Criteria:

1. It had received immunosuppressive drugs and cytotoxic therapy within the past 3 months more than 4 weeks;
2. It had received corticosteroids (prednisone or prednisolone) within the past 3 months more than 20mg/d for more than up to 4 weeks;
3. Acute or progressive glomerulonephritis patients;
4. Severe complications threat to life, such as severe infection;
5. Active hepatitis B and liver function test sustained abnormal;
6. Patients with malignant tumor or have a history of cancer, HIV infection, history of mental illness, acute central nervous system diseases, severe gastrointestinal diseases, prohibition of the use of hormone;
7. Abnormal glucose metabolism, fasting blood glucose over 6.2mmol/L;
8. Gravid or lactation woman;
9. Other clinical trials are being studied;
10. Merger with other serious disease and dysfunction of the organ.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate | changes from Baseline to 2, 4, 12, 24,36 and 48 weeks

SECONDARY OUTCOMES:
24-hour urinary protein excretion | changes from Baseline to 2, 4, 12, 24,36 and 48 weeks
serum creatinine | changes from Baseline to 2, 4, 12, 24,36 and 48 weeks
serum Lipid | Half-yearly
TCM syndrome score | changes from Baseline to 2, 4, 12, 24,36 and 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology,Longhua Hospital, Shanghai, China